CLINICAL TRIAL: NCT05745831
Title: Development and Validation of a Therapeutic Decision Aid in Less Active Ectopic Pregnancy
Brief Title: Development and Validation of a Therapeutic Decision Aid in Ectopic Pregnancy: GEUDECID Study
Acronym: GEUDECID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C22-51
Record Dates: First submitted 2023-02-01; First posted 2023-02-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2024-06

CONDITIONS: To Validate a Decision Aid for Ectopic Pregnancy
Keywords: decision aid; shared decision making; less active ectopic pregnancy; methotrexate; medical treatment; surgery

STUDY DESIGN:
Intervention Model Description: Prospective mulicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with a less active ectopic pregnancy using a therapeutic decision tool for treatment decision (Experimental): Women will have a therapeutic decision tool to help medical decision making and women and doctors will have to fill a questionnaire about the tool and the decision made
  Interventions: Other: Therapeutic decision tool

INTERVENTIONS:
Other: Therapeutic decision tool — A therapeutic decision tool will be used and its usefulness, comprehension and satisfaction will be evaluated

SUMMARY:
The aim's study is to validate a therapeutic aid in women with a less active ectopic pregnancy. A prospective recrutement of 100 women will be performed in 16 different hospitals in France. The decision aid will be used and a questionnaire about its usefulness, comprehension and satisfaction will be given to women and doctors.

DETAILED DESCRIPTION:
In less active ectopic pregnancy, two treatments are possible: a medical treatment using methotrexate or a surgical management.

A discret choice experiment study was performed to reveal women's preferences between these two options. In conclusion, calculated preferences are 47.5 and 52.5%, revealing a difficult choice for women. This study also lead to identify the main attributes important to make the choice. We were then able to create a therapeutic decision aid to help this shared decision.

This aid needs to be validated, following steps for validation. This study is the last step in women in situation of less active ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women who speak and read french
* Not opposed to participate to the research
* With a tubal ectopic pregnancy visible at sonography
* with an HCG rate under 10 000UI/ml

Exclusion Criteria:

* Cardiac activity present in the embryo
* Hemoperitoin
* Hemodynamic instability
* Spontaneous pelvic pain
* Contre indication to methotrexate
* Protected adult patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2023-10-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Validate acceptability of the therapeutic decision tool in women managed for less active ectopic tubal pregnancy. | One day
  Acceptability will be evaluated using a score from the Traditional Decisional Conflict Scale (DCS) translated in french. Women will fill it after the choice of the treatment and the realisation of it.

SECONDARY OUTCOMES:
Validate acceptability of the therapeutic decision tool in doctors who managed women for less active ectopic tubal pregnancy. | One day
  The same Traditional Decisional Conflict Scale (DCS) will be used in gynecologist who will managed the women
To evaluate satisfaction of women and of doctor in using the tool | One day
  A specific questionnaire using Likert scale will be used

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Service de gynécologie-obstétrique - Ch Montargis, Amilly
  - Service de Gynécologie-obstétrique - CHU Angers, Angers
  - Service de gynécologie-obstétrique - Hôpital Femme Mère Enfant, Bron
  - Service de gynécologie-obstétrique - CHU Caen, Caen
  - Service de Gynécologie-obstétrique - CHU Estaing, Clermont-Ferrand
  - Service Gynécologie - Hopital Bicêtre, Le Kremlin-Bicêtre
  - Service de gynécologie-obstétrique - CH Saint Vincent de Paul et Saint Philibert, Lille
  - Service de Gynécologie-obstétrique - Hopital Jeanne de Flandre, Lille
  - Service de gynécologie-obstétrique - Hopital Croix Rousse, Lyon
  - Service de gynécologie-obstétrique -CHU Arnaud De Villeneuve, Montpellier
  - Sevrice de gynécologie-obstétrique - CHU Nantes, Nantes
  - Service de Gynécologie-obstétrique - CHU Nîmes -, Nîmes
  - Service de gynécologie-obstétrique - CHU Rennes, Rennes
  - Service de gynécologie-obstétrique - CHU St Etienne, Saint-Etienne
  - Service de gynécologie-obstétrique - CHU Tours bretonneau, Tours

REFERENCES:
- [Result] Capmas P, Panjo H, Artignan J, Babelhadj A, Benoist I, Decouzon J, Jarrige C, Leglise M, Renoncet V, Pelletier-Fleury N. Women's preferences for less active ectopic pregnancy treatment: A discrete choice experiment. Eur J Obstet Gynecol Reprod Biol. 2024 Jan;292:175-181. doi: 10.1016/j.ejogrb.2023.11.032. Epub 2023 Nov 24. PMID 38035866